CLINICAL TRIAL: NCT00822783
Title: An Exploratory 16 Week, Double Blind, Placebo-Controlled Single Center Mechanistic Study to Determine the Effect of Rhumab-E25 on Phenotype and Function of IgE Mediated Antigen Presentation by Dendritic Cells in Subjects With Atopic Dermatitis.
Brief Title: Study to Determine the Effect of an Anti-IgE Agent on Inflammatory Cells in the Skin of Atopic Dermatitis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Other Study IDs: CIGE025A2412
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Atopic Dermatitis
Keywords: Serum IgE levels; inflammatory cells in the skin; inflammatory cells in the blood; IgE; IgE depletion; atopic dermatitis; atopic eczema; Omalizumab
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omalizumab (Active Comparator)
  Interventions: Drug: Omalizumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omalizumab
  Arms: Omalizumab
Drug: Placebo
  Arms: Placebo

SUMMARY:
Elevated levels of immunoglobuline E in blood are said to promote the occurence of atopic dermatitis; in fact, many patients with atopic dermatitis have high IgE levels. This study tried to explore whether the depletion of IgE from blood and skin might result in a change of immunological parameters and might alter the clinical course of the disease.

ELIGIBILITY:
Inclusion Criteria:

* aged between 12 and 60 years
* clinical diagnosis of AD (criteria of Hanifin and Rajka, 1980)
* serum IgE between 30 and 1,300 IU/ml
* at least one significantly positive RAST
* a positive skin prick test of the same specificity as the RAST
* an Investigator's Global Assessment Score of 2 or more at randomization
* stable AD, as defined as active AD (IGA 2 or more) for > 9 months per year
* signed informed consent.

Exclusion Criteria:

* pregnant or nursing females or women of childbearing potential who did not use a reliable contraceptive method
* treatment with omalizumab within the last 12 months before study treatment
* known hypersensitivity to any ingredients of omalizumab or omalizumab- related drugs
* elevated serum IgE levels for reasons other than atopy
* ongoing immunotherapy
* use of long-acting antihistamine astemizol within 3 months prior to visit1
* use of medium-acting antihistamines (e.g. loratadine, cetirizine) within 5 days prior to visit 1
* use of short-acting antihistamines (e.g. diphenhydramin, terfenadine) within 3 days prior to visit 1
* use of zafirlukast or other leukotriene receptor inhibitors and zileuton or other 5-lipoxygenase enzyme inhibitors within 3 days prior to visit 1
* use of phototherapy or systemic therapy that is known or suspected to have had an effect on AD within 1 month prior to first application of study medication
* treatment with topical therapy (other than hydrocortisone 1%) that is known or suspected to have had an effect on AD within 14 days prior to first application of study medication
* use of systemic steroids (oral, intravenous, including intraarticular and rectal) within one month prior to first application of study medication. (Patients on a stable maintenance dose of inhaled steroids were allowed to participate)
* use of systemic antibiotics within 2 weeks prior to first application of study medication
* use of tranquilizers, hypnotic agents or tricyclic antidepressants within 2 weeks prior to the start of the study
* immunocompromised patients or patients having a history of malignant disease
* concurrent skin diseases
* active bacterial, viral or fungal infections that required treatment with a prohibited medication
* a history of recurrent herpes simplex infection having active lesions at baseline
* tinea corporis / tinea cruris
* clinically significant laboratory abnormalities
* a history of noncompliance to medical regimens and patients who were considered potentially unreliable
* evidence of drug or alcohol abuse or other factors limiting ability to fully cooperate
* any condition or prior/continuing treatment which, in the opinion of the investigator, should have rendered the patient ineligible for the study.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2001-10; Study Completion 2003-04

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Immunology, Allergy and Infectious Diseases, Department of Dermatology, Medical University of Vienna, Austria., Vienna, Waehringer Guertel 18-20, Austria

REFERENCES:
- [Background] Lane JE, Cheyney JM, Lane TN, Kent DE, Cohen DJ. Treatment of recalcitrant atopic dermatitis with omalizumab. J Am Acad Dermatol. 2006 Jan;54(1):68-72. doi: 10.1016/j.jaad.2005.09.030. Epub 2005 Nov 28. PMID 16384758
- [Background] Krathen RA, Hsu S. Failure of omalizumab for treatment of severe adult atopic dermatitis. J Am Acad Dermatol. 2005 Aug;53(2):338-40. doi: 10.1016/j.jaad.2005.02.014. PMID 16021135
- [Background] Maurer D, Ebner C, Reininger B, Fiebiger E, Kraft D, Kinet JP, Stingl G. The high affinity IgE receptor (Fc epsilon RI) mediates IgE-dependent allergen presentation. J Immunol. 1995 Jun 15;154(12):6285-90. PMID 7759866
- [Background] Maurer D, Fiebiger E, Reininger B, Ebner C, Petzelbauer P, Shi GP, Chapman HA, Stingl G. Fc epsilon receptor I on dendritic cells delivers IgE-bound multivalent antigens into a cathepsin S-dependent pathway of MHC class II presentation. J Immunol. 1998 Sep 15;161(6):2731-9. PMID 9743330